CLINICAL TRIAL: NCT00792870
Title: Evaluation of the Shape Up Rhode Island Campaign: Study 4 Does Adding Behavioral Weight Control Information to Shape-Up Rhode Island Improve Outcomes?
Brief Title: Evaluation of the Shape Up Rhode Island Campaign
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Rena R. Wing, Professor, The Miriam Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 209707
Record Dates: First submitted 2008-11-14; First posted 2008-11-18 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Obesity
Keywords: Obesity; Weight loss; Internet
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SURI Enhanced (Experimental)
  Interventions: Behavioral: Evaluation of the Shape Up RI Campaign
- SURI Standard (Active Comparator)
  Interventions: Behavioral: Evaluation of the Shape Up RI Campaign

INTERVENTIONS:
Behavioral: Evaluation of the Shape Up RI Campaign — The SURI Standard group will receive all of the Shape-Up RI program materials plus an organized directory of useful websites related to healthy eating, exercise, and weight control. The SURI enhanced group will receive the standard Shape-Up RI program materials plus access to 12 behavioral weight loss lessons.

SUMMARY:
Obesity is a major health problem that has reached epidemic levels. Efforts are needed to develop cost-effective public health approaches for weight loss and maintenance. One such approach is to develop team-based programs that may motivate people to lose weight and/or increase their physical activity. One such program is entitled Shape-up Rhode Island (SURI). The purpose of this project is to evaluate the overall effectiveness of SURI and to test if a behavioral intervention can enhance the effectiveness of the original program. The current trial is investigating whether adding a behavioral intervention delivered online would enhance the outcomes of SURI participants.

DETAILED DESCRIPTION:
Background: Given the epidemic of obesity, approaches to weight loss that can be applied on a community, state, or national level are needed. This project is an ongoing evaluation of Shape Up Rhode Island (SURI) program, a state-wide Internet based program involving team-based competition to increase physical activity and achieve weight loss.

Aim: To enhance the effectiveness of SURI utilizing a minimal contact intervention delivered online.

Design: SURI 2008 participants were invited to join a research study focusing on weight loss. Interested participants were randomized to two groups including a SURI Enhanced (behavioral intervention presented in 12 weekly online presentations) or a SURI Standard group (group given a list of previously existing online resources to aid with weight loss).

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese
* Current participant in the Shape Up RI program weight loss competition

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Weight loss at the end of Shape Up RI | 3 months

SECONDARY OUTCOMES:
Weight loss maintenance 6 months after program completion | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rena R Wing, Ph.D., Principal Investigator — The Miriam Hospital
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States